CLINICAL TRIAL: NCT05206500
Title: Clinical Implication of Next Generation Sequencing of Urinary Bacteria in Patients With Low Colony Forming Units of Bacteria in Traditional Urine Culture
Brief Title: NextGen - Clinical Implication of Next Generation Sequencing
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00073565
Record Dates: First submitted 2022-01-07; First posted 2022-01-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Anti-Bacterial Agents; Ampicillin; Amoxicillin; Folic Acid Antagonists; Cephalosporins; Clindamycin; Fluoroquinolones; Fosfomycin; Linezolid; Metronidazole; Nitrofurantoin; Penicillins; Tetracyclines

STUDY DESIGN:
Intervention Model Description: Patients with Urinary Tract Infection (UTI) symptoms and Colony-forming Units (CFU) <10,000 have clinically significant UTIs. Characterizing the species of bacteria growing in low numbers and treating the patients based on bacterial sensitivity will help in resolving patients' symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Symptomatic Patients with low Colony Count (Other): Patients with positive urinalysis, symptomatic, and Urine Culture Colony Count <10,000 to be treated based on Next Generation Sequencing result.
  Interventions: Drug: Antibiotic; Device: Next Gen

INTERVENTIONS:
Drug: Antibiotic — FDA approved and marketed antibiotic treatment for the patients with UTI symptoms and CC >0 and <10,000
  Other Names: Ampicillin/Amoxicillin; Antifolates; Cephalosporins; Clindamycin; Extended spectrum penicillins; Fluoroquinolones; Fosfomycin; Linezolid; Metronidazole; Nitrofurantoin; Penicillins; Tetracyclines
Device: Next Gen — Next Generation Sequencing (NGS) is available to detect bacteria in urine based on bacterial genomes.

SUMMARY:
Recently more advanced techniques, including Polymerase Chain Reaction (PCR) and Next Generation Sequencing (NGS) are available to detect bacteria in urine based on bacterial genomes. Comparing to traditional culture, these techniques have more sensitivity and could potentially be of a great help in patients with Colony Count of less than 10,000 and more than zero.

DETAILED DESCRIPTION:
Bacterial sensitivity test for different antibiotics are the most important guide for treatment of patients with UTI. Unfortunately, for patients with less than 10,000 Colony Count (CC), usually no sensitivity test is done and there is not any guide for appropriate antibiotic therapy for this group.

ELIGIBILITY:
Inclusion Criteria:

* Female at least 18 years of age
* U/C (Urinary Culture) growth of <10,000 Colony-Forming Units (CFU)
* Understanding and acceptance of the need to return for all scheduled follow-up visits
* Able to give informed consent

Exclusion Criteria:

* Catheter in use (Foley or suprapubic or intermittent)
* Not able to provide clean midstream urine
* Antibiotic consumption in the past 2 weeks before signing the consent
* Pregnant or Planning to Conceive
* Incarcerated

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Next Generation Sequencing (NGS) Results (numbers of colony count (CC)) of Urinary Tract Infection (UTI) | Baseline
  NGS Ability to Detect Bacteria among patients with UTI Colony Count (CC) of Bacteria <10,000. Result Measure: NGS CC 100 to 10,000
Next Generation Sequencing (NGS) Results (numbers of colony count (CC)) of Urinary Tract Infection (UTI) | 3 Weeks Post-Treatment
  NGS Ability to Detect Bacteria among patients with UTI Colony Count (CC) of Bacteria <10,000, Result Measure: NGS CC 100 to 10,000

SECONDARY OUTCOMES:
Patient Improvement (King's Questionnaire Outcome measure) in UTI symptoms with CC <10,000 | Baseline
  NGS result focused antibiotic treatment and symptom outcome with the measurement of King's Questionnaire Outcome. Result Measure: Mild, Moderate, and Severe UTI symptoms in last 12 and 24 hours on 7 questions with no symptoms as "0", Mild as "1", Moderate as "2", and Severe as "3"
Patient Improvement (King's Questionnaire Outcome measure) in UTI symptoms with CC <10,000 | 3 Weeks Post-Treatment
  NGS result focused antibiotic treatment and symptom outcome with the measurement of King's Questionnaire Outcome. Result Measure: Mild, Moderate, and Severe UTI symptoms in last 12 and 24 hours on 7 questions with no symptoms as "0", Mild as "1", Moderate as "2", and Severe as "3"

CONTACTS AND LOCATIONS:
Overall Officials: Majid Mirzazadeh, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data are not planned to be shared. All subject related information will be available under the subject ID.